CLINICAL TRIAL: NCT05870852
Title: The Effectiveness of ESWT and PNF Techniques Added to ESWT in Individuals With Scleroderma With Calcinosis
Brief Title: Effectiveness of ESWT and PNF in Scleroderma With Calcinosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istanbul University (Other)
Collaborators: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Tugba Civi Karaaslan, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IstanbulC5
Record Dates: First submitted 2023-05-04; First posted 2023-05-23 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Scleroderma; Calcinosis Cutis
Keywords: scleroderma; ESWT; PNF techniques
MeSH Terms: conditions — Scleroderma, Diffuse; Calcinosis Cutis | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESWT (Experimental): All individuals who will participate in the study will be treated once a week for 4-5 minutes in total 3 times with ESWT. 2000 impulses will be applied on calcinosis with 2.4 bar pressure and 5.0 Hz frequency.
  Interventions: Device: Extracorporeal Shock Wave Therapy (ESWT)
- ESWT+PNF (Experimental): PNF stretching techniques will be applied in addition to ESWT. PNF stretching techniques: It will be done with isometric contraction for 10 seconds against maximum resistance. 8-10 repetitions will be done. A 10-second listening interval will be left for active relaxation of the patient between the applications. PNF application will be done by the physiotherapist once a week. You will be asked to do the PNF stretching exercises taught once daily as a home program.
  Interventions: Device: Extracorporeal Shock Wave Therapy (ESWT); Other: PNF

INTERVENTIONS:
Device: Extracorporeal Shock Wave Therapy (ESWT) — ESWT will be done once a week for 4-5 minutes in total 3 times with ESWT. 2000 impulses will be applied on calcinosis with 2.4 bar pressure and 5.0 Hz frequency.
Other: PNF — PNF stretching techniques: It will be done with isometric contraction for 10 seconds against maximum resistance. 8-10 repetitions will be done. A 10-second listening interval will be left for active relaxation of the patient between the applications. PNF application will be done by the physiotherapist once a week. You will be asked to do the PNF stretching exercises taught once daily as a home program.
  Arms: ESWT+PNF

SUMMARY:
Investigation of the effects of ESWT and PNF exercises added to ESWT on calcinosis in Ssc patients. Calcinosis cutis is a common, difficult-to-treat manifestation of systemic sclerosis associated with high morbidity. The aim of this study is to investigate the efficacy of ESWT therapy for calcinosis cutis in Ssc patients. The effects on grip strength, sleep, function and quality of life will be investigated.

DETAILED DESCRIPTION:
In Ssc patients, ESWT and PNF exercises that they take to ESWT should not be taken on calcinosis. Calcinosis cutis is a common, difficult-to-treat manifestation of disseminated systemic sclerosis with high morbidity. The effects on machine power, sleep, function and quality of life will be investigated. Evaluation Methods - Treatment ROM (with goniometer), second force (dynamometer), ultrasound (evaluation of calcinosis size), DASH (evaluation of ability to maintain upper extremity activities) , HAMIS (hand function test patient-specific functions assessment), Pitsburgh Sleep Quality Index (PUKI) - (Sleep assessment assessment), Pain assessment (with VAS), Health assessment questionnaire (SHAQ) (health status assessment) will be evaluated. As a result of the evaluation, two groups will be separated and one group will be ESWT, one group will be applied PNF stretching in addition to EWST. Treatment PNf Tension : 10 sec against max resistance. The time will be done with isometric contraction. 5 sec. It will wait for active circuit. 8-10 will be repeated. 10 seconds between applications. listening range will be left. PNF will be applied 3 times a week, once a week. ESWT: ESWT will be applied 3 times in total, 20 minutes once a week. 2000 impulses will be applied on calcinosis. The Patients will do the taught PNF exercises once a day as a home program. H1: PNF stretching exercises go on calcinosis when Ssc patients go to ESWT and ESWT. H2: ESWT and decreased to ESWT in Ssc patients PNF stretching exercises were not effective on calcinosis.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with SSc according to ACR/EULAR 2013 criteria
* Being diagnosed with Calcinosis by a physician
* Have the ability to adapt to exercises
* Stability of medical treatments

Exclusion Criteria:

* Being diagnosed with a known additional rheumatological or chronic disease
* Having a deformity that prevents doing the exercises
* Cognitive impairment
* Being pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-05-22 (Estimated); Primary Completion 2024-04-22 (Estimated); Study Completion 2024-05-22 (Estimated)

PRIMARY OUTCOMES:
Scleroderma Hand Mobility Test (HAMIS) | on the first day and three week change
  The hand function test developed for SSc patients will be used to assess patients' specific functions. The ability to use the hand in daily work and the limitation of movement will be evaluated. Finger movements, grasping, releasing, pronation, supination movements will be scored between 0-3. A lower total score of the scale indicates better functional activity.

SECONDARY OUTCOMES:
The Scleroderma Health Assessment Questionnaire (SHAQ) | on the first day and three week change
  The survey includes; Five visual analog scales questioning disease severity in general, as well as Raynaud's phenomenon, digital ulcer, gastrointestinal, and pulmonary respiratory symptoms. These questions are calculated separately and the score of each is between 0-3. The scale includes a 20-question Health Assessment Questionnaire (HAQ) that evaluates the functional competence level of the patient. This section includes fine motor movements of the upper extremity, locomotor activities of the lower extremity, and activities related to both the upper and lower extremities. The questions are scored between 0-3 (0=No difficulty and 3=Cannot). While scoring the sections, the highest score among the items that make up those 18 sections will be accepted as the section score. The score of each category will be summed and divided by 8, which is the total number of categories, to obtain the SHAQ score.
Arm, Shoulder and Hand Problems Questionnaire (DASH) | on the first day and three week change
  The ability of patients to perform certain upper extremity activities will be evaluated with a 30-item questionnaire. Patients will be asked to rate their level of difficulty with daily living on a five-point Likert scale. The calculation of the questionnaire, which can be used in any person with one or more upper extremity musculoskeletal disorders, is as follows: scoring formula = ([(sum of n answers)/n] -1). Higher scores indicate a higher level of disability and severity, while lower scores indicate a lower level of disability. The total score ranges from 0 (no disability) to 100 (most severe disability).
The Pittsburgh Sleep Quality Index (PSQI) | on the first day and three week change
  It is a sleep questionnaire that helps to evaluate sleep quality, amount of sleep, presence and severity of sleep disorder for the last month. There are 19 items in this scale and subjective sleep quality (C1), time to fall asleep (C2), sleep duration (C3), habitual sleep efficiency (C4), sleep disorders (C5), use of sleeping pills (C6) and daytime dysfunction ( It measures seven sub-components of sleep quality, including C7). The total PUKI score is obtained by summing the seven sub-scores and the total score is between 0-21. The PUKI total score clearly distinguishes good sleepers (PUKI total score ≤5) from poor sleepers (PUKI >5).
Visual Analog Scale (VAS) | on the first day and three week change
  The Pain Assessment will be evaluated with the visual analog scale (VAS). In order to be able to evaluate the pain subjectively, the individual will be asked to mark three different pain intensity levels in the joint with calcinosis on the pain scale evaluated out of 10: at rest, during activity and during sleep. The patient was asked to rate this scale (0: no pain, 10: severe pain) and determine a number accordingly for the severity of pain. Determining the pain level of the test by marking is an important advantage for ease of application.

CONTACTS AND LOCATIONS:
Overall Officials: TUGBA CIVI KARAASLAN, PhD, Principal Investigator — Istanbul University - Cerrahpasa